CLINICAL TRIAL: NCT05106309
Title: A Phase 1, Open-label Trial to Evaluate the Pharmacokinetics of CVL-231 Following Single Oral Administration of Modified- and Immediate-release Formulations Under Fasted and Fed Conditions in Healthy Participants
Brief Title: Pharmacokinetics of CVL-231 Following Single Oral Administration of Modified- and Immediate-release Formulations in Fasted and Fed Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cerevel Therapeutics, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CVL-231-1004
Record Dates: First submitted 2021-11-01; First posted 2021-11-03 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Healthy Volunteer; Schizophrenia Spectrum and Other Psychotic Disorders; Mental Disorders
MeSH Terms: conditions — Schizophrenia; Schizophrenia Spectrum and Other Psychotic Disorders; Mental Disorders

STUDY DESIGN:
Intervention Model Description: Part A is an open-label, randomized, 4-period, 4-sequence, crossover design to investigate the PK, relative bioavailability, safety, and tolerability of single doses of CVL-231 IR/MR formulations in healthy participants. The following treatments, administered under fasted conditions are: 1) 10mg CVL-231 as IR formulation, 2) 30mg CVL-231 as slow release MR formulation, 3) 30mg CVL-231 as medium release MR formulation, 4) 30mg CVL-231 as fast release MR formulation.
  Part B is an open-label, randomized, 2-period, 2-sequence, crossover design to investigate the effect of food on CVL-231 PK following a single dose of the CVL-231 MR formulation in healthy participants. After completion of Part A, a target release formulation (MR formulation with acceptable PK characteristics) may be selected and effect of food on CVL-231 PK from the target release formulation may be evaluated. Based on Part A data, if a target release formulation cannot be selected, Part B of the trial may be canceled.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part A: Single doses of CVL-231 IR/MR formulations in healthy participants under fasted conditions (Experimental): Oral Dose
  Interventions: Drug: 10 mg CVL-231 as IR formulation; Drug: 30 mg CVL-231 as slow-release MR formulation; Drug: 30 mg CVL-231 as medium release MR formulation; Drug: 30 mg CVL-231 as fast release MR formulation
- Part B: Single doses of CVL-231 target release formulation under fasted and fed conditions (Experimental): Oral Dose
  Interventions: Drug: 30 mg CVL-231 Target Release, Fasted; Drug: 30 mg CVL-231 Target Release, Fed

INTERVENTIONS:
Drug: 10 mg CVL-231 as IR formulation — Tablets
  Arms: Part A: Single doses of CVL-231 IR/MR formulations in healthy participants under fasted conditions
Drug: 30 mg CVL-231 as slow-release MR formulation — Capsules
  Arms: Part A: Single doses of CVL-231 IR/MR formulations in healthy participants under fasted conditions
Drug: 30 mg CVL-231 as medium release MR formulation — Capsules
  Arms: Part A: Single doses of CVL-231 IR/MR formulations in healthy participants under fasted conditions
Drug: 30 mg CVL-231 as fast release MR formulation — Capsules
  Arms: Part A: Single doses of CVL-231 IR/MR formulations in healthy participants under fasted conditions
Drug: 30 mg CVL-231 Target Release, Fasted — Capsules
  Arms: Part B: Single doses of CVL-231 target release formulation under fasted and fed conditions
Drug: 30 mg CVL-231 Target Release, Fed — Capsules
  Arms: Part B: Single doses of CVL-231 target release formulation under fasted and fed conditions

SUMMARY:
A 2-part, crossover design, open-label treatment trial with 4 periods, 4 sequences (Part A) to evaluate MR formulations of CVL-231 and a 2 periods, 2 sequences (Part B) to understand effect of food on CVL-231 exposures from an MR formulation.

DETAILED DESCRIPTION:
CVL-231 is a muscarinic acetylcholine receptor (mAChR) activator that selectively binds to the M4 muscarinic receptor subtype (M4 mAChR) and is being developed for treatment of psychosis in schizophrenia. Part A of this 2-part trial will investigate the PK of CVL-231 in healthy participants following a single oral dose of CVL-231 as 3 modified-release (MR) formulations with different release rates and an immediate-release (IR) formulation under fasted conditions. Upon selection of an MR formulation with appropriate PK characteristics, the effect of food on the PK of CVL-231 and its metabolite following single oral doses of the selected MR formulation may be evaluated in Part B.

ELIGIBILITY:
Inclusion Criteria:

1. Women of nonchildbearing potential and men 18 to 55 years, inclusive.
2. Healthy as determined by medical evaluation, including medical and psychiatric history, physical and neurological examinations, ECG, vital sign measurements, and laboratory test results, as evaluated by the investigator.
3. Body mass index of 18.5 to 30.0 kg/m2 and a total body weight >50 kg (110 lbs).
4. Sexually active men with a pregnant or a nonpregnant partner of childbearing potential must agree to comply with protocol contraception requirements during treatment and through 7 days post dose. In addition, male participants should not donate sperm for a minimum of 7 days following the last dose of IMP.
5. Capable of giving signed informed consent.
6. Ability, in the opinion of the investigator, to understand the nature of the trial and comply with protocol requirements.

Exclusion Criteria:

1. Current history of significant cardiovascular, pulmonary, gastrointestinal, renal, hepatic, metabolic, endocrine, hematological, immunological, or neurological disease that, in the opinion of the investigator or medical monitor, could compromise either participant safety or the results of the trial.
2. Current or past personal or family history of any psychiatric disorder as classified by DSM-5 criteria.
3. Epilepsy or a history of seizures except for a single seizure episode, eg, a childhood febrile seizure, a seizure related to trauma or alcohol withdrawal, or an unexplained loss of consciousness.
4. History of moderate to severe substance or alcohol-use disorder (excluding caffeine) within 12 months prior to signing the ICF.
5. Serious risk of suicide in the opinion of the investigator
6. Receipt of SARS-CoV2 vaccine or booster within 28 days of dosing with CVL-231, or plan to receive SARS-CoV2 vaccination or booster from Screening through 5 days after last dose of CVL-231.
7. Have recently been diagnosed with symptomatic COVID-19 or test positive for COVID-19 within 30 days prior to signing the ICF.
8. Either of the following:

   * History of HIV, hepatitis B, or hepatitis C infection
   * Positive result for HIV antibody, hepatitis B surface antigen, hepatitis B core antibody, or hepatitis C antibody
9. Positive drug screen for illicit drugs or a positive test for alcohol
10. 12-lead ECG demonstrating pre-defined abnormalities at Screening and Day -1 based on local evaluation.
11. Abnormal clinical laboratory tests or vital sign measurements at the Screening Visit and at Day -1 (check-in) for each period
12. Known to be allergic or hypersensitive to the IMP or any of its components.
13. Participation in any clinical trial within 90 days prior to signing the ICF.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2021-12-29 (Actual); Primary Completion 2022-02-24 (Actual); Study Completion 2022-02-24 (Actual)

PRIMARY OUTCOMES:
Primary Part A & B: Peak Plasma Concentration (Cmax) for CVL-231 and Metabolite (CV-0000364) | Up to 72 Hours in each period
Primary Part A & B: Time to Maximum Concentration (Tmax) for CVL-231 and Metabolite (CV-0000364) | Up to 72 Hours in each period
Primary Part A & B: Time prior to the first measurable (non-zero) concentration (Tlag) for CVL-231 and Metabolite (CV-0000364) | Up to 72 Hours in each period
Primary Part A & B: Area under the plasma concentration-time curve from time 0 to the last measurable time point (AUClast) for CVL-231 and Metabolite (CV-0000364) | Up to 72 Hours in each period
Primary Part A & B: Area under the plasma concentration-time curve from time zero to infinity (AUCinf) for CVL-231 and Metabolite (CV-0000364) | Up to 72 Hours in each period
Primary Part A & B: Elimination half-life (t½) for CVL-231 and Metabolite (CV-0000364) | Up to 72 Hours in each period
Primary Part A only: Dose normalized Cmax, derived by Cmax divided by the dose administered (Cmax/D) for CVL-231 and Metabolite (CV-0000364) | Up to 72 Hours in each period
Primary Part A only: Dose normalized AUClast, derived by AUClast divided by the dose administered (AUClast/D) for CVL-231 and Metabolite (CV-0000364) | Up to 72 Hours in each period
Primary Part A only: Dose normalized AUCinf, derived by AUCinf divided by the dose administered (AUCinf/D) for CVL-231 and Metabolite (CV-0000364) | Up to 72 Hours in each period

SECONDARY OUTCOMES:
Secondary: Incidence and Severity of Treatment Emergent Adverse Events (TEAEs) | Up to Day 14
Secondary: Incidence of clinically significant changes in electrocardiogram (ECG) results | Up to 72 Hours in each period
  Assessment of clinically significant changes in QT intervals measured by 12-lead ECG recording after the participant has been supine and at rest for at least 3 minutes.
Secondary: Incidence of clinically significant changes in clinical laboratory results | Up to 72 Hours in each period
Secondary: Incidence of clinically significant changes in vital sign measurements | Up to 72 Hours in each period
  Assessment of clinically significant changes in vital signs including temperature, systolic and diastolic blood pressure, and heart rate.
Secondary: Incidence of clinically significant changes in physical and neurological examination results | Up to 72 Hours in each period
Secondary: Clinically significant findings in suicidality assessed using the Columbia Suicide-Severity Rating Scale (C-SSRS) | Up to 72 Hours in each period
  The C-SSRS rates an individual's degree of suicidal ideation (SI) on a scale, ranging from "wish to be dead" to "active suicidal ideation with specific plan and intent." The scale identifies SI severity and intensity, which may be indicative of an individual's intent to commit suicide. C-SSRS SI severity subscale ranges from 0 (no SI) to 5 (active SI with plan and intent).

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Leoni, MD, MBA, Study Director — Cerevel Therapeutics, LLC
Locations (1):
- Celerion Inc., Tempe, Arizona, United States